CLINICAL TRIAL: NCT00000922
Title: A Randomized, Open-Label Study of the Long-Term Effectiveness of Three Initial Highly Active Antiretroviral Therapy (HAART) Strategies in HAART-Niave, HIV-Infected Persons
Brief Title: A Study to Evaluate the Long-Term Effectiveness of Three Anti-HIV Drug Regimens in HIV Infected Patients Who Have Never Been Exposed to Highly Active Antiretroviral Therapy (HAART)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPCRA 058; 11611 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; abacavir; Nelfinavir; efavirenz; Nevirapine; Lamivudine; Stavudine; Didanosine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Abacavir sulfate
Drug: Nelfinavir mesylate
Drug: Efavirenz
Drug: Nevirapine
Drug: Lamivudine
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to determine whether it is better to start an anti-HIV regimen containing a protease inhibitor (PI), a non-nucleoside reverse transcriptase inhibitor (NNRTI), or a PI in combination with an NNRTI. This study will also examine which treatment regimen is best as a first treatment for HIV infection.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) regimens containing PIs, NNRTIs, or nucleoside reverse transcriptase inhibitors (NRTIs) have been shown to slow disease progression. However, the long-term consequences of initial therapy with a PI, an NNRTI, or both a PI and an NNRTI are not yet known, nor is the impact on future anti-HIV treatment regimens. Patients who experience virologic failure on a particular HAART regimen typically have not been studied for subsequent response to other HAART regimens. It is possible that a regimen which is initially the most potent may not be optimal if it limits the effectiveness of subsequent anti-HIV treatment regimens.

Patients will be randomized to one of three HAART treatment arms:

* Arm 1 participants will receive one or two PIs plus two NRTIs.
* Arm 2 participants will receive one NNRTI plus two NRTIs.
* Arm 3 participants will receive one or two PIs plus an NNRTI plus one or two NRTIs.

Before randomization to a treatment arm, patients will be given the option of preselecting the drugs they will use or allowing randomization to study-specified drugs. The study-specified PIs will be indinavir (IDV), nelfinavir (NFV), or two PIs of patient and doctor choice. The study-specified NNRTIs will be nevirapine (NVP) or efavirenz (EFV). The study-specified NRTIs will be abacavir (ABC) plus lamivudine (3TC) or didanosine (ddI) plus stavudine (d4T).

The study sites will provide ABC, 3TC, ddI, or d4T to all patients who are assigned to take these medications. All other anti-HIV drugs for initial and subsequent treatment regimens are obtained by clinician prescription. At Months 1 and 4 and then every 4 months thereafter, patients will receive a medical history update, physical exam, and questionnaire. Blood samples will also be drawn to measure CD4 cell count, viral load, and genotypic antiretroviral resistance. Changes in treatment regimens may occur at any time.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Agree to practice abstinence or to use barrier methods of birth control during the study
* Are at least 13 years old or have signed informed consent from legal guardian for patients between the ages of 13 and 18

Exclusion Criteria:

* Have ever taken any anti-HIV drugs
* Are unable to complete the study for any reason
* Pregnancy
* Breastfeeding
* Any condition that, in the investigator's opinion, may interfere with the study

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1710
Dates: Primary Completion 2003-01 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Change in CD4 count from baseline to the average of all readings obtained at the regular follow-up visits beginning at Month 32
time to disease progression, death, or CD4 count less than 200 cells/mm3 at the 4 Month visit for those patients with a baseline CD4 cell count of more than or equal to 200 cells/mm3

CONTACTS AND LOCATIONS:
Overall Officials: Rodger D. MacArthur, MD, Study Chair — University Health Center, Wayne State University; Richard Novak, MD, Study Chair — University of Illinois at Chicago
Locations (17):
- United States (17):
  - Community Consortium / UCSF, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Yale Univ School of Medicine / AIDS Program, New Haven, Connecticut
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Wayne State Univ - WSU/DMC / Univ Hlth Ctr, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners in Research / New Mexico, Albuquerque, New Mexico
  - Harlem AIDS Treatment Grp / Harlem Hosp Ctr, New York, New York
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Univ TX Health Science Ctr, Houston, Texas
  - Richmond AIDS Consortium / Div of Infect Diseases, Richmond, Virginia

REFERENCES:
- [Background] Moyle GJ, DeJesus E, Cahn P, Castillo SA, Zhao H, Gordon DN, Craig C, Scott TR; Ziagen Once-Daily in Antiretroviral Combination Therapy (CNA30021) Study Team. Abacavir once or twice daily combined with once-daily lamivudine and efavirenz for the treatment of antiretroviral-naive HIV-infected adults: results of the Ziagen Once Daily in Antiretroviral Combination Study. J Acquir Immune Defic Syndr. 2005 Apr 1;38(4):417-25. doi: 10.1097/01.qai.0000147521.34369.c9. PMID 15764958
- [Background] Ribera E, Rodriguez-Pardo D, Rubio M, Soler A, Pedrol E, Blanco JL, Gonzalez A, Crespo M, Falco V, Ocana I, Deig E, Miro JM, Pahissa A. Efficacy and safety of once-daily combination therapy with didanosine, lamivudine and nevirapine in antiretroviral-naive HIV-infected patients. Antivir Ther. 2005;10(5):605-14. PMID 16152754
- [Background] Shlay JC, Visnegarwala F, Bartsch G, Wang J, Peng G, El-Sadr WM, Gibert C, Kotler D, Grunfeld C, Raghavan S; Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA). Body composition and metabolic changes in antiretroviral-naive patients randomized to didanosine and stavudine vs. abacavir and lamivudine. J Acquir Immune Defic Syndr. 2005 Feb 1;38(2):147-55. doi: 10.1097/01.qai.0000143599.64234.15. PMID 15671799
- [Result] MacArthur RD, Chen L, Mayers DL, Besch CL, Novak R, van den Berg-Wolf M, Yurik T, Peng G, Schmetter B, Brizz B, Abrams D; CPCRA 058 FIRST Trial Study Team. The rationale and design of the CPCRA (Terry Beirn Community Programs for Clinical Research on AIDS) 058 FIRST (Flexible Initial Retrovirus Suppressive Therapies) trial. Control Clin Trials. 2001 Apr;22(2):176-90. doi: 10.1016/s0197-2456(01)00111-8. PMID 11306155
- [Result] Tedaldi EM, Absalon J, Thomas AJ, Shlay JC, van den Berg-Wolf M. Ethnicity, race, and gender. Differences in serious adverse events among participants in an antiretroviral initiation trial: results of CPCRA 058 (FIRST Study). J Acquir Immune Defic Syndr. 2008 Apr 1;47(4):441-8. doi: 10.1097/QAI.0b013e3181609da8. PMID 18176329
- [Result] van den Berg-Wolf M, Hullsiek KH, Peng G, Kozal MJ, Novak RM, Chen L, Crane LR, Macarthur RD; CPCRA 058 Study Team, the Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA), and The International Network for Strategic Initiative in Global HIV Trials (INSIGHT). Virologic, immunologic, clinical, safety, and resistance outcomes from a long-term comparison of efavirenz-based versus nevirapine-based antiretroviral regimens as initial therapy in HIV-1-infected persons. HIV Clin Trials. 2008 Sep-Oct;9(5):324-36. doi: 10.1310/hct0905-324. PMID 18977721
- [Result] MacArthur RD, Novak RM, Peng G, Chen L, Xiang Y, Hullsiek KH, Kozal MJ, van den Berg-Wolf M, Henely C, Schmetter B, Dehlinger M; CPCRA 058 Study Team; Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA). A comparison of three highly active antiretroviral treatment strategies consisting of non-nucleoside reverse transcriptase inhibitors, protease inhibitors, or both in the presence of nucleoside reverse transcriptase inhibitors as initial therapy (CPCRA 058 FIRST Study): a long-term randomised trial. Lancet. 2006 Dec 16;368(9553):2125-35. doi: 10.1016/S0140-6736(06)69861-9. PMID 17174704